CLINICAL TRIAL: NCT05361122
Title: Prevention of Developmental Delay and Xylitol (PDDaX) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Gregory C. Valentine, MD MED FAAP, Assistant Professor: Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00015305
Record Dates: First submitted 2022-04-27; First posted 2022-05-04 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Prematurity; Neurodevelopmental Disorders
Keywords: Xylitol; Oral Health; Pregnancy; Prematurity
MeSH Terms: conditions — Premature Birth; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: We will enroll 1000 children aged 4-8 years of age. n=500 will be former term children and additional n=500 will be former preterm children. Half in each group (n=250) will be gestationally xylitol-exposed, and the other half (n=250) will not be xylitol-exposed.
Who Masked: Care Provider
Masking Description: Psychologists and dentists will be blinded to the treatment status (xylitol or no xylitol use during pregnancy) of the mothers of the pediatric subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Xylitol-exposed formerly term children (Experimental): n=250 formerly term children born during the PPaX trial who were born to gravidae in the interventional arm (received xylitol chewing gum but had access to a dentist and received prenatal counseling)
  Interventions: Dietary Supplement: Maternal Use of Xylitol Chewing Gum During Pregnancy
- Non xylitol-exposed formerly term children (Active Comparator): n=250 formerly term children born during the PPaX trial who were born to gravidae in the active comparator arm (no xylitol chewing gum but had access to a dentist and received prenatal counseling)
  Interventions: Dietary Supplement: No Maternal Xylitol Chewing Gum Use During Pregnancy
- Xylitol-exposed formerly preterm children (Experimental): n=250 formerly preterm children born during the PPaX trial who were born to gravidae in the interventional arm (received xylitol chewing gum but had access to a dentist and received prenatal counseling)
  Interventions: Dietary Supplement: Maternal Use of Xylitol Chewing Gum During Pregnancy
- Non xylitol-exposed formerly preterm children (Active Comparator): n=250 formerly preterm children born during the PPaX trial who were born to gravidae in the active comparator arm (no xylitol chewing gum but had access to a dentist and received prenatal counseling)
  Interventions: Dietary Supplement: No Maternal Xylitol Chewing Gum Use During Pregnancy

INTERVENTIONS:
Dietary Supplement: Maternal Use of Xylitol Chewing Gum During Pregnancy — There are no current interventions within this follow-up study. However, the mothers enrolled in the parent PPaX trial received xylitol-containing chewing gum (1 gram per stick of gum and instructed to chew 1-2 sticks of gum twice daily for a total dose of 2-4 grams/day of xylitol throughout pregnancy starting pre-conception or at <20 weeks gestation).
  Arms: Xylitol-exposed formerly preterm children; Xylitol-exposed formerly term children
Dietary Supplement: No Maternal Xylitol Chewing Gum Use During Pregnancy — There are no current interventions within this follow-up study. Children born to mothers who received access to a dentist and prenatal education (oral health, prevention of preterm birth) are in the active comparator group
  Arms: Non xylitol-exposed formerly preterm children; Non xylitol-exposed formerly term children

SUMMARY:
The goals of this study are to: evaluate and validate the low-cost, transportable, easily-administered Malawi Developmental Assessment Tool (MDAT) for neurodevelopmental assessment of children aged 4-8 years old in Malawi, as compared to the gold-standard yet more cumbersome and costly Kaufman Assessment Battery for Children-II (KABC-II) among (1) n=500 formerly preterm children and (2) n=500 formerly term children.

Additionally, we will evaluate the effects of gestational xylitol exposure compared to a lack of gestational xylitol exposure on neurodevelopmental outcomes of children aged 4-8 years old in Malawi through the following four neurodevelopmental tests: (3) KABC-II (cognitive outcomes), (4) EF Touch (executive functions), (5) Strengths and Difficulties Questionnaire (social-emotional outcomes), and (6) MDAT (motor and cognitive outcomes).

The researchers will leverage subjects who completed the parent Prevention of Prematurity and Xylitol Trial, which enrolled 10069 pregnant individuals in Malawi and demonstrated a significant 24% reduction in incidence of preterm birth and low birthweight offspring in gravidae who chewed xylitol-containing chewing gum compared to those who did not. By ensuring that these offspring did not have higher rates of neurodevelopmental impairment, the study will promote promising multi-center international and domestic trial evaluating the impact of xylitol-containing chewing gum use and optimal dosage during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Child born during the PPaX trial
* Enrollment age between 4-8 years old
* Parental or legal guardian consent obtained
* Willing to undergo 3 neurodevelopmental tests
* Willing to travel to BCMF for neurodevelopmental assessment
* Assent by the pediatric subject for participation in the study

Exclusion Criteria:

* Parent or legal guardian cognitively unable to provide consent
* Child unwilling to provide assent to participate in the study

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Validation of the MDAT in Former Preterm Children | 1 month (1-2 clinic visits)
  compared to the KABC-II
Validation of the MDAT in Former Term Children | 1 month (1-2 clinic visits)
  compared to the KABC-II
KABC-II mental processing index | 1 month (1-2 clinic visits)
  In n=500 former term and n=500 former preterm children aged 4-8 years old with half of each being gestationally xylitol exposed vs not exposed
EF Touch composite score | 1 month (1-2 clinic visits)
  In n=500 former term and n=500 former preterm children aged 4-8 years old with half of each being gestationally xylitol exposed vs not exposed
SDQ composite | 1 month (1-2 clinic visits)
  In n=500 former term and n=500 former preterm children aged 4-8 years old with half of each being gestationally xylitol exposed vs not exposed
MDAT composite neurodevelopmental outcome | 1 month (1-2 clinic visits)
  In n=500 former term and n=500 former preterm children aged 4-8 years old with half of each being gestationally xylitol exposed vs not exposed

SECONDARY OUTCOMES:
Incidence of cognitive delay per specific KABC-II subdomain | 1 month (1-2 clinic visits)
  sequential processing (working memory), simultaneous processing (visual processing), planning ability (fluid reasoning), and learning ability (long-term memory and retrieval)
Incidence of executive function delay per specific EF Touch subdomains | 1 month (1-2 clinic visits)
  processing speed ("Bubbles"), visual spatial working memory ability ("Farmer"), working memory ("Pick the Picture" and "Houses"), inhibitory motor control ("Pig", "Silly Sounds Game", and "Arrows"), and Flexible thinking ("Something's the Same")
Incidence of social-emotional delay per specific SDQ subdomains | 1 month (1-2 clinic visits)
  Emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior
Incidence of neurodevelopmental delay as per MDAT subdomains | 1 month (1-2 clinic visits)
  Gross motor, fine motor, social, and language

CONTACTS AND LOCATIONS:
Overall Officials: Greg Valentine, MD, Principal Investigator — University of Washington
Locations (1):
- Baylor College of Medicine Children's Foundation-Malawi, Lilongwe, Malawi

REFERENCES:
- [Derived] Valentine GC, Collett B, Wallie S, Mhango J, Engmann C, Sullivan E, Seferovic M, Willoughby M, Shayo B, Walson JL, Milgrom P, Aagaard K, Juul SE. The Prevention of Developmental Delay and Xylitol (PDDaX) trial: study protocol of a nested cohort follow-up from the PPaX (Prevention of Prematurity and Xylitol) trial examining neurodevelopmental outcomes among offspring at 4-8 years of age in Malawi. Trials. 2025 Nov 14;26(1):506. doi: 10.1186/s13063-025-09204-y. PMID 41239527